CLINICAL TRIAL: NCT05203432
Title: The Effect and Safety of Red Light Intervention on Myopic Progression of Myopic Children: Randomized Clinical Trial
Brief Title: Red Light Intervention on Myopic Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21Y11910000
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Light Intervention (Experimental): Repeated Low-Level Red-Light Therapy
  Interventions: Device: Red Light Intervention
- Low concentration atropine (Active Comparator): 0.01% atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Device: Red Light Intervention — Repeated Low-Level Red-Light Therapy
  Arms: Red Light Intervention
Drug: Atropine — 0.01% atropine
  Arms: Low concentration atropine

SUMMARY:
To explore the effectiveness of using repeated low-level red-light therapy to slow myopia progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrolment: 6-12 years;
2. At least one eye with spherical equivalent refractions (SERs): -1.00 to -5.00 diopters (D), and stigmatism of 1.50 D or less;
3. Anisometropia of 1.5 D or less;
4. The BCVA of distant vision is at least 0.8;
5. Myopia progressed more than 0.5D in the past year;
6. Have normal thinking and language communication skills, and be able to actively cooperate with the treatment as required;
7. Written informed consent of guardian and child.

Exclusion Criteria:

1. Strabismus, amblyopia or other ocular abnormalities;
2. Other systemic abnormalities;
3. Prior treatment of myopia control in 6 months, e.g. drugs, orthokeratology, progressive addition lenses, bifocal lenses, etc in either eye;
4. Atropine allergy;
5. Other situations that not suitable for participating in the trial as judged by the researcher.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of axial length | at least 1 year
  AL was measured as the distance from the anterior corneal surface to the retinal pigment epithelium (RPE) using IOLMaster

SECONDARY OUTCOMES:
Change of spherical equivalent | at least 1 year
  Spherical equivalent as measured by cycloplegia autorefraction
Change of choroidal thickness | at least 1 year
  Choroidal thickness will be measured using SS-OCT
Change of uncorrected visual acuity | at least 1 year
  Uncorrected visual acuity (UCVA) will be measured using a mounted and illuminated E chart of the Early Treatment Diabetic Retinopathy study (ETDRS) charts.

CONTACTS AND LOCATIONS:
Overall Officials: Jiannan Huang, Principal Investigator — Shanghai Eye Disease Prevention and Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, China